CLINICAL TRIAL: NCT00828217
Title: ACTIVHOP: Adapted Physical Activity, Health-related Quality of Life and Satisfaction With Care in Hospitalized Children; a Randomized Controlled Study
Brief Title: Adapted Physical Activity, Health-related Quality of Life and Satisfaction With Care in Hospitalized Children
Acronym: ACTIVHOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Nancy (Other); Association pour la promotion du sport chez l'enfant malade (APSEM) (Unknown)
Responsible Party: Chastagner Pascal, MD, PhD, University Hospital of Nancy
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AC-2008-HO
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Hospitalization
Keywords: adapted physical activity; hospital; health-related quality of life; satisfaction with care; child; adolescent; randomized controlled trial; physical activity; quality of life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- with APA (Experimental): Children have adapted physical activity during their hospitalization
  Interventions: Other: adapted physical activity
- without APA (No Intervention): Children don't have adapted physical activity during their hospitalization

INTERVENTIONS:
Other: adapted physical activity — one session of adapted physical activity per day (30 minutes each session), during the whole stay at the hospital
  Arms: with APA

SUMMARY:
The aim of this study is to assess the efficacy of adapted physical activity intervention on health-related quality of life and satisfaction with care in hospitalized children and adolescents.

This is a randomized controlled study. The hypothesis is that children practicing adapted physical activity during their hospitalization present a higher health-related quality of life and satisfaction with care than those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Length of hospital stay (more than 3 days)
* Children or parents able to understand and read French
* No medical contra-indications to physical activity
* Children hospitalized in 3 specific departments at Nancy Children's Hospital:

  * Médecine Infantile 1 et 3(paediatrics)
  * Médecine Infantile 2 (haematology-oncology, immunology department)
  * Chirurgie orthopédique et Brûlés (orthopaedic surgery and Burned)
* Children and parents being agree to participate in the study

Exclusion Criteria:

* No written informed consent
* Children hospitalized less than 3 days
* Medical contra-indication to physical activity
* Children already included in that study (former hospitalization)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 312 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
health-related quality of life measurement | 2 points: on the first and last day of hospitalization

SECONDARY OUTCOMES:
satisfaction with care measurement | 1 point: 15 days after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Chastagner, MD, PhD, Principal Investigator — University Hospital of Nancy, Children's Hospital; Serge Briançon, Pr, Study Chair — Nancy-University, Paul Verlaine Metz University, Paris Descartes University, EA4360 Apemac, Nancy, France; Anne Vuillemin, PhD, Study Chair — Nancy-University, Paul Verlaine Metz University, Paris Descartes University, EA4360 Apemac, Nancy, France; Aline Herbinet, PhD, Study Chair — APSEM
Locations (1):
- University Hospital, Children's Hospital, Vandœuvre-lès-Nancy, France